CLINICAL TRIAL: NCT01734434
Title: A Multicenter, Observational Study to Identify Factors That Influence Access of Pregnant Women and Their Infants to Their Local Healthcare Systems
Brief Title: Study to Identify Factors Influencing Access of Pregnant Women and Their Infants to Local Healthcare Systems
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V98_15OB
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2017-07

CONDITIONS: Pregnancy, Newborn Health
Keywords: Health care access, Pregnant women

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: 24 weeks or more of gestation

SUMMARY:
This study collected information regarding the factors that might influence access of pregnant women to the local healthcare system. The main visits of the study screened & enrollment, delivery and 90 day infant follow-up. Data were collected mainly from questionnaires administered to pregnant women at these visits. The questionnaires contained the following standard questions which were asked at each visit, in addition to some visit-specific questions related to delivery and health status of infants up to 90 days of age. The standard questions related to the following aspects:

* Logistics of transportation to the study site (type, time it takes, cost incurred)
* Accessibility to a telephone/cell phone
* Provisions of alternative child care during site visits if there are other children under the subject's care

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with gestational age of greater than or equal to 24 weeks at the time of enrollment
2. Subject / subject's parents or a legal representative who has given written consent after the nature of the study has been explained according to local regulatory requirements
3. Pregnant women of gestational age between 28 weeks and 34 weeks 6/7 days

Exclusion Criteria:

None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women of gestational age 24 weeks or more
Sampling Method: Probability Sample
Enrollment: 3243 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (10):
- Dominican Republic (2):
  - Centro Sanitario de Santo Domingo, Santo Domingo
  - Maternidad Nuestra Senora de La Altagracia, Santo Domingo
- CISM Manhica Health Research Centre, Manhiça, Mozambique
- Panama (3):
  - Policentro Juan Diaz, Panama City
  - Policentro Parque Lefevre, Panama City
  - Policlínica JJ Vallarino, Panama City
- South Africa (4):
  - Children's Infectious Diseases Clinical Research Unit, Cape Town
  - Setshaba Research Centre, Gauteng
  - Synexus Research Centre, Gauteng
  - Respiratory and Meningeal Pathogens Research Unit, Soweto, Johannesburg

REFERENCES:
- [Background] WHO. Antenatal care in developing countries. Promises, achievements and missed opportunities. An analysis of trends, levels and differentials, 1990-2001. Geneva: 2003.
- [Background] Assembly UNG. A world fit for children. Outcome document of the Special Session on Children. New York: 2002.
- [Background] Qazi SA, Stoll BJ. Neonatal sepsis: a major global public health challenge. Pediatr Infect Dis J. 2009 Jan;28(1 Suppl):S1-2. doi: 10.1097/INF.0b013e31819587a9. No abstract available. PMID 19106756
- [Derived] Madhi SA, Rivera LM, Saez-Llorens X, Menendez C, Carrim-Ganey N, Cotton MF, Katzman D, Luttig MM, Candelario R, Baker S, Roychoudhury M. Factors influencing access of pregnant women and their infants to their local healthcare system: a prospective, multi-centre, observational study. BMC Pregnancy Childbirth. 2018 Jan 15;18(1):29. doi: 10.1186/s12884-017-1655-3. PMID 29334920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Dominican Republic, Panama, Mozambique, and South Africa.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Maternal Subjects (Dominican Republic): Pregnant women who were enrolled in Dominican Republic.
- Maternal Subjects (Panama): Pregnant women who were enrolled in Panama.
- Maternal Subjects (South Africa): Pregnant women who were enrolled in South Africa.
- Maternal Subjects (Mozambique): Pregnant women who were enrolled in Mozambique.
Period: Overall Study
Arm/Group | Maternal Subjects (Dominican Republic) | Maternal Subjects (Panama) | Maternal Subjects (South Africa) | Maternal Subjects (Mozambique)
Started | 500 | 500 | 1992 | 251
Completed | 490 | 488 | 1863 | 228
Not Completed | 10 | 12 | 129 | 23
Not completed — Death Infant | 3 | 1 | 17 | 5
Not completed — Lost to Follow-up | 2 | 9 | 67 | 11
Not completed — No Live Birth | 1 | 2 | 32 | 6
Not completed — Withdrawal by Subject | 4 | 0 | 8 | 1
Not completed — Signed Adult Version of Consent Form | 0 | 0 | 1 | 0
Not completed — Subject Not Reachable | 0 | 0 | 1 | 0
Not completed — Treatment Defaulter | 0 | 0 | 1 | 0
Not completed — Wrong Version of Consent Form Signed | 0 | 0 | 1 | 0
Not completed — 17 Yr Old Subject Signed Consent form | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data was analysed on Full analysis set (FAS) population-All subjects in the all enrolled set who provided data after enrollment related to delivery, logistics or medical outcomes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Subjects (Dominican Republic) | Maternal Subjects (Panama) | Maternal Subjects (South Africa) | Maternal Subjects (Mozambique) | Total
Number analyzed (Participants) | 500 | 500 | 1989 | 251 | 3240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.49 (5.28) | 25.08 (5.65) | 27.05 (6.05) | 25.01 (6.26) | 26.19 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 500 | 500 | 1989 | 251 | 3240
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Delivering at a Study Site.
Description: The percentage of subjects who delivered at the study site relative to the number of enrolled subjects was calculated
Time Frame: Baseline until average of 24 weeks
Population: Analysis was done on Full analysis set (FAS)-All subjects in the All Enrolled Set who provided data after enrollment related to delivery, logistics or medical outcomes.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Maternal Subjects (Dominican Republic) | Maternal Subjects (Panama) | Maternal Subjects (South Africa) | Maternal Subjects (Mozambique)
Number analyzed (Participants) | 500 | 500 | 1989 | 251
Percentages of subjects
  Subjects with known delivery information | 99.20 [97.96 to 99.78] | 100 [99.26 to 100] | 99.65 [99.28 to 99.86] | 100 [98.54 to 100]
  Study site delivery | 68.55 [64.26 to 72.61] | 74.40 [70.34 to 78.17] | 56.66 [54.44 to 58.86] | 86.85 [82.03 to 90.77]

2. Primary Outcome: Percentage of Subjects Delivering at a Non-study Site.
Description: The percentage of subjects who delivered at a non-study site relative to the number of enrolled subjects was calculated.
Time Frame: Baseline until average of 24 weeks
Population: Analysis was done on FAS.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Maternal Subjects (Dominican Republic) | Maternal Subjects (Panama) | Maternal Subjects (South Africa) | Maternal Subjects (Mozambique)
Number analyzed (Participants) | 500 | 500 | 1989 | 251
Percentages of subjects
  Subjects with known delivery information | 99.20 [97.96 to 99.78] | 100 [99.26 to 100] | 99.65 [99.28 to 99.86] | 100 [98.54 to 100]
  Non-study healthcare facility | 30.85 [26.81 to 35.12] | 24.60 [20.88 to 28.62] | 41.32 [39.14 to 43.53] | 7.97 [4.93 to 12.04]
  Home | 0 [0 to 0] | 0.40 [0.05 to 1.44] | 0.76 [0.42 to 1.25] | 2.79 [1.13 to 5.66]
  Other | 0 [0 to 0] | 0 [0 to 0] | 0.50 [0.24 to 0.93] | 0.40 [0.01 to 2.20]
  Unknown | 0.60 [0.12 to 1.76] | 0.60 [0.12 to 1.74] | 0.76 [0.42 to 1.25] | 1.99 [0.65 to 4.59]

3. Secondary Outcome: Number of Infants Born Live, Reported Sick and Brought to a Study or Non-study Health Care Facility Site.
Description: The number of infants born live, reported sick and brought to a study or non-study health care facility site by the maternal subjects over the period of 90 days after delivery was calculated.
Time Frame: Delivery to Day 90 post-delivery (Infant follow-up)
Population: Analysis was done on the FAS
Measure: Number; unit: participants
Groups:
- Maternal Subjects(Dominican Republic): pregnant women who were enrolled in Dominican Republic.
- Maternal Subjects(Panama): pregnant women who were enrolled in Panama.
- Maternal Subjects(Mozambique): pregnant women who were enrolled in Mozambique.
Arm/Group | Maternal Subjects(Dominican Republic) | Maternal Subjects(Panama) | Maternal Subjects (South Africa) | Maternal Subjects(Mozambique)
Number analyzed (Participants) | 493 | 498 | 1966 | 242
participants
  Live births at discharge | 493 | 498 | 1966 | 242
  Infants reported sick | 58 | 81 | 74 | 5
  Infants brought to health care facility-study site | 54 | 147 | 27 | 51

4. Secondary Outcome: Number of Infants Brought to Study Site During Infant Follow up (90 Days Post-delivery)
Description: The number of infants who were brought by the maternal subjects to a study site for 90-day infant follow-up visit relative to the number of live birth deliveries.
Time Frame: Delivery to Day 90 post-delivery (Infant follow-up)
Population: Analysis was performed on the FAS.
Measure: Number; unit: participants
Groups:
- Infants (Dominican Republic): Infants born to pregnant women who were enrolled in Dominican Republic, brought to study site for 90-day follow up.
- Infants (Panama): Infants born to pregnant women who were enrolled in Panama, brought to study site for 90-day follow up.
- Infants (South Africa): Infants born to pregnant women who were enrolled in South Africa, brought to study site for 90-day follow up.
- Infants (Mozambique): Infants born to pregnant women who were enrolled in Mozambique, brought to study site for 90-day follow up.
Arm/Group | Infants (Dominican Republic) | Infants (Panama) | Infants (South Africa) | Infants (Mozambique)
Number analyzed (Participants) | 493 | 498 | 1966 | 242
participants | 479 | 333 | 1163 | 146

ADVERSE EVENTS:
Description: Adverse event data were not collected.
Arm/Group | Maternal Subjects (Dominican Republic) | Maternal Subjects (Panama) | Maternal Subjects (South Africa) | Maternal Subjects (Mozambique)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days